CLINICAL TRIAL: NCT03525028
Title: Multicenter, Randomized, Controlled Clinical Trial Research Evaluating the Use of Combination Therapy of Glucocorticoids and Metformin to Decrease Glucocorticoids Side Effects in Patients With Autoimmune Uveitis
Brief Title: A Clinical Trial of Metformin to Decrease Glucocorticoids Side Effects in Patients With Autoimmune Uveitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University (Other)
Collaborators: Peking Union Medical College Hospital (Other); Peking University First Hospital (Other); Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiaomin Zhang, Director of the Tianjin Medical University Eye Institute，archiater, Tianjin Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017KY-06
Record Dates: First submitted 2018-04-14; First posted 2018-05-15 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Uveitis; Metformin; Glucocorticoid
MeSH Terms: conditions — Uveitis | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin group (Experimental): Oral metformin 500 mg once daily for first week, 500 mg twice daily for next 23 weeks. The follow-up treatment according to the participants' condition.
  Interventions: Drug: Metformin
- Placebo group (Placebo Comparator): Oral placebo 500 mg once daily for first week, 500 mg twice daily for next 23 weeks. The follow-up treatment according to the participants' condition.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — The investigators assumed that the combination therapy of metformin and glucocorticoids can decrease glucocorticoids side effects and synergia the anti-inflammatory and immune inhibitory effect of glucocorticoids. So the investigators use metformin in the experimental group.
  Arms: Metformin group
Drug: Placebo — The investigators use placebo in the control group.
  Arms: Placebo group

SUMMARY:
This project is designed to evaluating the use of combination therapy of glucocorticoid and metformin to decrease glucocorticoid side effects in participants with autoimmune uveitis.This study also aims to evaluate the anti-inflammatory and immunosuppressive effects of combination therapy.

DETAILED DESCRIPTION:
Approval of the study was obtained from the hospital's ethical committee. The study design and methodology followed the tenets of Declaration of Helsinki. All participants were provided with written informed consent and received a thorough explanation of the study design, aims, and the side effect of metformin. This is a multicenter, randomized, controlled clinical trial research. According to 1:1 ratio, all participants are randomly divided into two groups, the metformin group and placebo group.

According to the fasting blood glucose (FBG), triglycerides (TG),total cholesterol (TC) and body mass index (BMI), the investigators compared experimental group with control group to evaluate whether the use of combination therapy of glucocorticoid and metformin decrease glucocorticoid side effects in participants with autoimmune uveitis.

According to best corrected visual acuity (BCVA), anterior chamber and vitreous inflammation, fluorescence fundus angiography (FFA), electroretinogram (ERG) and so on, the investigators evaluate the anti-inflammatory and immunosuppressive effects of metformin in treatment of autoimmune uveitis.

ELIGIBILITY:
Inclusion Criteria:

1. Attending Tianjin Medical University Eye Hospital, ophthalmology department of Peking Union Medical College Hospital, ophthalmology department of Peking University First Hospital and Zhongshan Ophthalmic Center Sun Yat-sen University from January 2018 to January 2022.
2. Chronic and non-infectious autoimmune uveitis with systemic glucocorticoids treatment (Initiation dosage ≥ 1 mg/kg/d or ≥ 50 mg/d).
3. FBG < 6.1 mmol/L, HbAlc<6.O%, TC <6.2 mmol/L(240 mg／d1) and TG <2.3 mmol/L(200 mg／dl).
4. All genders, age ≥ 18 years old.
5. Ready for systemic glucocorticoids treatment.
6. Willing to follow all study requirements and sign the informed consent.
7. Without history of cancer and serious systemic diseases.

Exclusion Criteria:

1. Participate in other clinical trials within the preceding one years
2. Planning ophthalmologic surgery over the next three months.
3. With other sight-threatening diseases except cataract, such as glaucoma, diabetic retinopathy, retinal detachment, and so on.
4. Taking or will take immunosuppressants which affecting glycometabolism and lipid metabolism except methotrexate,mycophenolate and azathioprine.
5. Any known history of a serious infection (e.g., HIV, hepatitis, pneumonia, syphilis or tuberculosis).
6. Any known history of diabetes mellitus, severe hepatic, renal or heart disease.
7. Any known history of drug addiction, drug abuse and malignant tumor.
8. Presence of a transplanted solid organ.
9. Pregnant women and nursing mothers.
10. Any known history of mental disorders.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of abnormal metabolic indexes | 24 weeks
  The assessments of abnormal metabolic indexes include any of these outcome measures: FBG≥6.1 mmol/L, TC≥6.2 mmol/L (240 mg/d1), TG≥2.3 mmol/L (200 mg/dl) or BMI increased 1 kg/m^2 than before in the process of follow-up twice in a row.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaorong Li, M.D., Study Director — Tianjin Medical University Eye Hospital
Locations (1):
- Tianjin Medical University Eye Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The study protocol,statistical analysis plan,informed consent form and clinical study report are to be shared with other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will become available starting 6 months after publication.
Access Criteria: The study protocol,statistical analysis plan,informed consent form and clinical study report are to be shared with other researchers.

REFERENCES:
- [Background] Del Barco S, Vazquez-Martin A, Cufi S, Oliveras-Ferraros C, Bosch-Barrera J, Joven J, Martin-Castillo B, Menendez JA. Metformin: multi-faceted protection against cancer. Oncotarget. 2011 Dec;2(12):896-917. doi: 10.18632/oncotarget.387. PMID 22203527
- [Result] Hoes JN, van der Goes MC, van Raalte DH, van der Zijl NJ, den Uyl D, Lems WF, Lafeber FP, Jacobs JW, Welsing PM, Diamant M, Bijlsma JW. Glucose tolerance, insulin sensitivity and beta-cell function in patients with rheumatoid arthritis treated with or without low-to-medium dose glucocorticoids. Ann Rheum Dis. 2011 Nov;70(11):1887-94. doi: 10.1136/ard.2011.151464. Epub 2011 Sep 10. PMID 21908880
- [Result] den Uyl D, van Raalte DH, Nurmohamed MT, Lems WF, Bijlsma JW, Hoes JN, Dijkmans BA, Diamant M. Metabolic effects of high-dose prednisolone treatment in early rheumatoid arthritis: balance between diabetogenic effects and inflammation reduction. Arthritis Rheum. 2012 Mar;64(3):639-46. doi: 10.1002/art.33378. PMID 21953589
- [Result] Schacke H, Docke WD, Asadullah K. Mechanisms involved in the side effects of glucocorticoids. Pharmacol Ther. 2002 Oct;96(1):23-43. doi: 10.1016/s0163-7258(02)00297-8. PMID 12441176
- [Result] Oray M, Abu Samra K, Ebrahimiadib N, Meese H, Foster CS. Long-term side effects of glucocorticoids. Expert Opin Drug Saf. 2016;15(4):457-65. doi: 10.1517/14740338.2016.1140743. Epub 2016 Feb 6. PMID 26789102
- [Result] Gulliford MC, Charlton J, Latinovic R. Risk of diabetes associated with prescribed glucocorticoids in a large population. Diabetes Care. 2006 Dec;29(12):2728-9. doi: 10.2337/dc06-1499. No abstract available. PMID 17130214
- [Result] Perez A, Jansen-Chaparro S, Saigi I, Bernal-Lopez MR, Minambres I, Gomez-Huelgas R. Glucocorticoid-induced hyperglycemia. J Diabetes. 2014 Jan;6(1):9-20. doi: 10.1111/1753-0407.12090. Epub 2013 Oct 29. PMID 24103089
- [Result] Pasieka AM, Rafacho A. Impact of Glucocorticoid Excess on Glucose Tolerance: Clinical and Preclinical Evidence. Metabolites. 2016 Aug 3;6(3):24. doi: 10.3390/metabo6030024. PMID 27527232
- [Result] Kahn BB, Alquier T, Carling D, Hardie DG. AMP-activated protein kinase: ancient energy gauge provides clues to modern understanding of metabolism. Cell Metab. 2005 Jan;1(1):15-25. doi: 10.1016/j.cmet.2004.12.003. PMID 16054041
- [Result] Jeon SM. Regulation and function of AMPK in physiology and diseases. Exp Mol Med. 2016 Jul 15;48(7):e245. doi: 10.1038/emm.2016.81. PMID 27416781